CLINICAL TRIAL: NCT04453553
Title: COVID-19 in Vitro Diagnostic Near-patient Testing in Care Environments Using a Cluster Randomised Open-label Trial Design in an East London Care Home Population
Brief Title: CICERO- A Care Home Study of COVID-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in government policy on testing
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 285524
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: COVID
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: randomised cluster trial of care homes
Masking Description: No masking will be used as the study arms have different testing patterns
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Screening for COVID-19 via nasopharyngeal swab taken at day 0 and 14
  Interventions: Diagnostic Test: Nasopharyngeal swab and main laboratory
- Near Patient Testing (Experimental): Screening for COVID-19 via nasopharyngeal swab taken at day 0 and 14, with the addition of daily nasal swabs tested via rapid test system
  Interventions: Diagnostic Test: Q16 testing

INTERVENTIONS:
Diagnostic Test: Q16 testing — Nasal swab tested on a rapid near patient device
  Arms: Near Patient Testing
Diagnostic Test: Nasopharyngeal swab and main laboratory — Standard of care testing
  Arms: Standard of care

SUMMARY:
The primary objective of the study is to determine whether, at 21 days, care homes that implemented near-patient daily testing have a lower rate of confirmed CoV-2 infections than care homes following the DHSC standard of care testing of symptomatic residents.

DETAILED DESCRIPTION:
Accurate, rapid, near-patient testing systems, such as q16+CoV-2, allow for daily routine testing of residents, and of staff and visitors prior to entering the care home.

Daily CoV-2 PCR testing with high analytical sensitivity (e.g., 2 copies per 8 µl sample) may detect infected residents and visitors before clinical symptoms are apparent. Earlier detection may lead to earlier implementation of the UK standard of care protocol for Infection prevention and control measures, thereby preventing the asymptomatic infected individuals from introducing and/or transmitting CoV-2 within the care home. This should reduce the transmission by:

Preventing the introduction of the virus into care homes from external visitors e.g., GPs (Inward transmission) Preventing the spread of the virus within care homes and preventing cluster development (internal transmission) Preventing the outward spread of the virus from within care homes by infection of external visitors (Outward transmission)

ELIGIBILITY:
Inclusion Criteria:

* Persons resident or requiring access to the care home
* Capable of giving written informed consent, or if appropriate, having an acceptable individual capable of giving consent on the participant's behalf.

Exclusion Criteria:

* Persons not providing informed consent or withdrawing consent at any time during the study.
* Persons requiring urgent and immediate access to the care home, for example medical staff attending emergency visits.
* Persons unable to provide nasal or oropharyngeal swabs for medical reasons.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
CoV-2 Infection after 21 days | 21 days
  The cumulative number of confirmed cases of CoV-2 infection after 21 days, measured by PCR detection of CoV-2, within the care home residents, staff and visitors

SECONDARY OUTCOMES:
CoV-2 Infection after 14 days | 14 days
  The cumulative number of confirmed cases of CoV-2 infection after 14 days, measured by PCR detection of CoV-2, within the care home residents, staff and visitors.
Cases of suspected or confirmed CoV-2 infection | 14 days
  The cumulative number of suspected or confirmed cases of CoV-2 infection after 14 days, within the care home residents, staff and visitors.
Hospitalisation and death | 21 days and 40 days
  The cumulative number of confirmed COVID-19-related hospitalisations and deaths of care home residents, staff and visitors after 21 and 40 days.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Martin, Study Chair — Queen Mary University London
Locations (1):
- Queen Mary University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Public Health England. Outbreaks in Care Homes in England. Cumulative data to 17th May 2020
- [Background] University of Cambridge, MRC Biostatistics Unit. Nowcasting and Forecasting of COVID-19
- [Background] Comas-Herrera A and Zalakain J. Mortality associated with COVID-19 outbreaks in care homes: early international evidence. 12th April 2020
- [Background] McMichael TM, Currie DW, Clark S, Pogosjans S, Kay M, Schwartz NG, Lewis J, Baer A, Kawakami V, Lukoff MD, Ferro J, Brostrom-Smith C, Rea TD, Sayre MR, Riedo FX, Russell D, Hiatt B, Montgomery P, Rao AK, Chow EJ, Tobolowsky F, Hughes MJ, Bardossy AC, Oakley LP, Jacobs JR, Stone ND, Reddy SC, Jernigan JA, Honein MA, Clark TA, Duchin JS; Public Health-Seattle and King County, EvergreenHealth, and CDC COVID-19 Investigation Team. Epidemiology of Covid-19 in a Long-Term Care Facility in King County, Washington. N Engl J Med. 2020 May 21;382(21):2005-2011. doi: 10.1056/NEJMoa2005412. Epub 2020 Mar 27. PMID 32220208
- [Background] Kimball A, Hatfield KM, Arons M, James A, Taylor J, Spicer K, Bardossy AC, Oakley LP, Tanwar S, Chisty Z, Bell JM, Methner M, Harney J, Jacobs JR, Carlson CM, McLaughlin HP, Stone N, Clark S, Brostrom-Smith C, Page LC, Kay M, Lewis J, Russell D, Hiatt B, Gant J, Duchin JS, Clark TA, Honein MA, Reddy SC, Jernigan JA; Public Health - Seattle & King County; CDC COVID-19 Investigation Team. Asymptomatic and Presymptomatic SARS-CoV-2 Infections in Residents of a Long-Term Care Skilled Nursing Facility - King County, Washington, March 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 3;69(13):377-381. doi: 10.15585/mmwr.mm6913e1. PMID 32240128
- [Background] Roxby AC, Greninger AL, Hatfield KM, Lynch JB, Dellit TH, James A, Taylor J, Page LC, Kimball A, Arons M, Schieve LA, Munanga A, Stone N, Jernigan JA, Reddy SC, Lewis J, Cohen SA, Jerome KR, Duchin JS, Neme S. Detection of SARS-CoV-2 Among Residents and Staff Members of an Independent and Assisted Living Community for Older Adults - Seattle, Washington, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 10;69(14):416-418. doi: 10.15585/mmwr.mm6914e2. PMID 32271726
- [Background] World Health Organisation (WHO). Coronavirus disease 2019 (COVID-19) situation report 73. 2020
- [Background] Mizumoto K, Kagaya K, Zarebski A, Chowell G. Estimating the asymptomatic proportion of coronavirus disease 2019 (COVID-19) cases on board the Diamond Princess cruise ship, Yokohama, Japan, 2020. Euro Surveill. 2020 Mar;25(10):2000180. doi: 10.2807/1560-7917.ES.2020.25.10.2000180. PMID 32183930
- [Background] Sheridan C. Fast, portable tests come online to curb coronavirus pandemic. Nat Biotechnol. 2020 May;38(5):515-518. doi: 10.1038/d41587-020-00010-2. No abstract available. PMID 32203294
- [Background] Department of Health & Social Care. COVID-19: Our Action Plan for Adult Social Care. 15th April 2020
- [Background] He X, Lau EHY, Wu P, Deng X, Wang J, Hao X, Lau YC, Wong JY, Guan Y, Tan X, Mo X, Chen Y, Liao B, Chen W, Hu F, Zhang Q, Zhong M, Wu Y, Zhao L, Zhang F, Cowling BJ, Li F, Leung GM. Temporal dynamics in viral shedding and transmissibility of COVID-19. Nat Med. 2020 May;26(5):672-675. doi: 10.1038/s41591-020-0869-5. Epub 2020 Apr 15. PMID 32296168
- [Background] Foundation for Innovative New Diagnostics. SARS-CoV-2 Molecular Assay Evaluation: Results
- [Background] Primerdesign™ Ltd. Primerdesign Ltd COVID-19 genesig® Real-Time PCR assay. Instructions for Use. Issue 1.01. 20th March 2020. Available at: https://www.fda.gov/media/136309/download (page 21)
- [Background] Ip DKM, Lau LLH, Chan KH, Fang VJ, Leung GM, Peiris MJS, Cowling BJ. The Dynamic Relationship Between Clinical Symptomatology and Viral Shedding in Naturally Acquired Seasonal and Pandemic Influenza Virus Infections. Clin Infect Dis. 2016 Feb 15;62(4):431-437. doi: 10.1093/cid/civ909. Epub 2015 Oct 30. PMID 26518469
- [Background] NHS, PHE, DHSC and CQC. Admission and Care of Patients during COVID-19 Incident in a Care Home. 2nd April 2020. Version 1.